CLINICAL TRIAL: NCT03542591
Title: Supplementation of Critical Nutrients in a Plant-based Diet as Assessed by Experts in Nutrition - a Cross-sectional Survey
Brief Title: Supplementation of Critical Nutrients in a Plant-based Diet
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: VegMed2018
Record Dates: First submitted 2018-04-20; First posted 2018-05-31 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Deficiency, Vitamin; Vegan's Anemia (Vitamin B12 Deficiency); Deficiencies Micronutrient
MeSH Terms: conditions — Avitaminosis; Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants of the VegMed congress (Berlin, April 2018)
  Interventions: Other: Questionnaire on the topic "Supplementation of critical nutrients in a plant-based diet"

INTERVENTIONS:
Other: Questionnaire on the topic "Supplementation of critical nutrients in a plant-based diet" — No active intervention, only survey as mentioned above.

SUMMARY:
500 participants of the vegan/vegetarian congress VegMed are to be included, which should answer once (cross-sectional study) a medicine socio-behaviorist questionnaire on the topic "supplementation of critical nutrients in a plant-based diet" at the VegMed congress on 21/04/2018. The aim of the study is to understand how experts in this field behave and whether actions taken follow official recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the VegMed congress (Berlin, April 2018)
* Expertise of the respondent in the field of nutritional medicine
* Presence during the oral education to participate in the survey

Exclusion Criteria:

N/A

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Participants of the VegMed congress (Berlin, April 2018)
  * Expertise of the respondent in the field of nutritional medicine
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-04-21 (Actual)

PRIMARY OUTCOMES:
Assessment of critical nutrients in vegan diet | 21st April 2018
  Cross-sectional survey

SECONDARY OUTCOMES:
Supplementation of critical nutrients in a vegan diet | 21st April 2018
  Cross-sectional survey
Recommendations for patients by the experts | 21st April 2018
  Cross-sectional survey

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, Germany